CLINICAL TRIAL: NCT04890262
Title: Prospective, Non-interventional, Observational Study in Patients With IBD Receiving IV or SC Vedolizumab Therapy to Observe Route of Administration Choices and Outcomes (VARIETY-AUT)
Brief Title: A Study of Vedolizumab in Adults With Ulcerative Colitis (UC) or Crohn's Disease (CD) in Real-World Practice
Acronym: VARIETY-AUT
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: Vedolizumab-4035
Record Dates: First submitted 2021-05-13; First posted 2021-05-18 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Inflammatory Bowel Diseases; Crohns Disease; Colitis, Ulcerative
Keywords: Drug Therapy
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease; Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants With Inflammatory Bowel Disease (IBD): Participants diagnosed with moderately to severely active IBD (UC or CD) who are currently ongoing vedolizumab intravenous (IV) treatment in line with current Summary of Product Characteristics (SmPC) or local prescribing information with the option to switch to vedolizumab subcutaneous (SC) treatment, will be observed prospectively for 24 months.

SUMMARY:
Vedolizumab is a medicine that helps to reduce symptoms of IBD and the associated inflammation in the digestive system for participants with ulcerative colitis or Crohn's disease.

In this study, participants with ulcerative colitis or Crohn's disease will be treated with vedolizumab according to their clinic's standard practice. Participants will receive vedolizumab as either an infusion or an injection just under the skin (subcutaneous). The main aim of the study is to observe real-world treatment patterns in participants treated with vedolizumab.

The study sponsor will not be involved in how participants are treated but will provide instructions on how the clinics will record what happens during the study.

DETAILED DESCRIPTION:
This is a non-interventional, prospective study of participants with moderately to severely active IBD (UC or CD) who are initiating or currently ongoing induction or maintenance treatment with vedolizumab in the real world setting.

The study will enroll approximately 100 participants. The data will be collected prospectively at the study sites and will be recorded into electronic case report forms (e-CRFs). All the participants will be assigned to a single observational cohort:

* Participants with IBD

This multi-center study will be conducted in Austria at specialized gastroenterology centers. The overall duration of the study will be 24 months. Data will be collected at baseline, at 3 months after induction, and every 6 months after induction, and at the time of switch, discontinuation and/or at routine follow-up visits up to 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. Has moderately to severely active IBD (UC or CD), initiating or ongoing IV induction treatment with vedolizumab in accordance with the current SmPC at baseline OR IBD participants receiving ongoing/maintenance IV vedolizumab treatment, with the option to switch to SC vedolizumab maintenance treatment.

Exclusion Criteria:

1. Prior history of intolerability, hypersensitivity, or other contraindications (active severe infections such as tuberculosis, sepsis, cytomegalovirus, listeriosis, and opportunistic infections such as Progressive Multifocal Leukoencephalopathy) to vedolizumab therapy as defined in the current SmPC.
2. Current or planned participation in an interventional clinical trial for CD or UC.
3. Cognitive incapacity, unwillingness or language barriers precluding adequate understanding or cooperation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult participants with moderately to severely active UC or CD receiving vedolizumab treatment in accordance with the approved SmPC.
Sampling Method: Non-Probability Sample
Enrollment: 99 (Actual)
Dates: Start 2021-08-18 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants Persisting on Treatment With Vedolizumab IV Compared to Participants With Treatment Change up to 12 Months | Baseline up to 12 months
Time to any Treatment Change | Baseline up to 24 months
Number of Participants With Reason for Treatment Change | Baseline up to 24 months
Number of Participants With Change in Vedolizumab Dosing Frequency | Baseline up to 24 months
Number of Participants Who Discontinued Vedolizumab Treatment | Baseline up to 24 months
Number of Participants Who Changed to Another Treatment | Baseline up to 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (7):
- Austria (7):
  - Medizinische Universitat Graz, Graz
  - Medizinische Universitat Innsbruck, Innsbruck
  - JKU Linz, Linz
  - Krankenhaus der Barmherzigen Bruder, Saint Veit/Glan
  - Darmpraxis Salzburg, Salzburg
  - Medizinische Universitat Wien, Vienna
  - Klinikum Wels-Grieskirchen GmbH, Wels

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information on the study, click here/on this link. — https://clinicaltrials.takeda.com/study-detail/60a50c041f1122001e30a7db